CLINICAL TRIAL: NCT01595438
Title: A Phase III, Randomized, Multicenter, Double-Blind, Double Dummy, Parallel Group, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime Avibactam (CAZ-AVI, Formerly CAZ104) Versus Doripenem Followed by Appropriate Oral Therapy in the Treatment of Complicated Urinary Tract Infections, Including Acute Pyelonephritis, With a Gram Negative Pathogen in Hospitalized Adults
Brief Title: Ceftazidime-Avibactam Compared With Doripenem Followed by Oral Therapy for Hospitalized Adults With Complicated UTIs (Urinary Tract Infections)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4280C00002; 2011-005721-43
Record Dates: First submitted 2012-04-27; First posted 2012-05-10 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Complicated Urinary Tract Infection (cUTI) Including Acute Pyelonephritis
Keywords: Ceftazidime, Avibactam, Doripenem, Ciprofloxacin, sulfamethoxazole/trimethoprim, Anti-Infective Agents, Complicated Urinary Tract Infection,Acute Pyelonephritis
MeSH Terms: interventions — avibactam, ceftazidime drug combination; Doripenem; Ciprofloxacin; Sulfamethoxazole; Trimethoprim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ceftazidime - Avibactam ( CAZ-AVI) (Experimental): IV treatment
  Interventions: Drug: Ceftazidime - Avibactam ( CAZ-AVI); Drug: Either switch to oral therapy: 500 mg of Ciprofloxacin (oral); Drug: or switch to oral therapy: 800 mg/160 mg of sulfamethoxazole/trimethoprim (oral)
- Doripenem (Active Comparator): IV treatment
  Interventions: Drug: Doripenem; Drug: Either switch to oral therapy: 500 mg of Ciprofloxacin (oral); Drug: or switch to oral therapy: 800 mg/160 mg of sulfamethoxazole/trimethoprim (oral)

INTERVENTIONS:
Drug: Ceftazidime - Avibactam ( CAZ-AVI) — Ceftazidime 2000 mg and 500 mg of avibactam. Patients randomized to receive CAZ-AVI will receive an infusion of CAZ-AVI (2000 mg ceftazidime and 500 mg avibactam) every 8 hours administered by intravenous (IV) infusion in a volume of 100 mL at a constant rate over 120 minutes
  Arms: Ceftazidime - Avibactam ( CAZ-AVI)
Drug: Doripenem — 500 mg of Doripenem. Patients randomized to receive Doripenem will receive an infusion of Doripenem 500 mg every 8 hours administered by intravenous (IV) infusion in a volume of 100 mL at a constant rate over 60 minutes
  Arms: Doripenem
Drug: Either switch to oral therapy: 500 mg of Ciprofloxacin (oral) — Patients are eligible for oral switch after receiving 5 full days of IV therapy and have met protocol specified criteria for clinical improvement
Drug: or switch to oral therapy: 800 mg/160 mg of sulfamethoxazole/trimethoprim (oral) — Patients are eligible for oral switch after receiving 5 full days of IV therapy and have met protocol specified criteria for clinical improvement

SUMMARY:
The purpose of this study is to evaluate the effects of Ceftazidime Avibactam compared to Doripenem for treating hospitalized patients with complicated urinary tract infections, including acute pyelonephritis

DETAILED DESCRIPTION:
A Phase III, Randomized, Multicenter, Double-Blind, Double Dummy, Parallel Group, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime Avibactam (CAZ-AVI, formerly CAZ104) Versus Doripenem Followed by Appropriate Oral Therapy in the Treatment of Complicated Urinary Tract Infections, Including Acute Pyelonephritis, With a Gram Negative Pathogen in Hospitalized Adults

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years of age inclusive
* Female patients can participate if they are surgically sterile or completed menopause or females capable of having children and agree not to attempt pregnancy while receiving IV study therapy and for a period of 7 days after
* Has pyuria with >/= 10 WBCs (white blood cell) and has a positive urine culture within 48 hours of enrollment containing >/=10 to the fifth CFU (colony forming unit ) /ml of a recognized uropathogen known to be susceptible to IV study therapy (CAZ-AVI and doripenem)
* Demonstrates either acute pyelonephritis or complicated lower UTI without pyelonephritis.

Exclusion Criteria:

* Urine pathogen is a Gram-positive pathogen or a uropathogen resistant to CAZ-AVI or doripenem
* Patient's urine culture at study entry isolates more than 2 microorganisms regardless of colony count or patient has a confirmed fungal UTI
* Patient is receiving hemodialysis or peritoneal dialysis or had a renal transplant
* Patient is immunocompromised
* Patient is considered unlikely to survive the 6- to 8-week study period or has a rapidly progressive or terminal illness including septic shock which is associated with a high risk of mortality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MBBS, MRCP, Study Director — AstraZeneca
Locations (80):
- United States (3):
  - Research Site, Sylmar, California
  - Research Site, Royal Oak, Michigan
  - Research Site, Lima, Ohio
- Argentina (4):
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Santa Fe
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Campinas/SP
  - Research Site, Salvador
  - Research Site, São José Do Rio Preto - SP
  - Research Site, São Paulo
  - Research Site, Vila Clementino
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
- Research Site, Zagreb, Croatia
- Czechia (2):
  - Research Site, Kyjov
  - Research Site, Opava
- Germany (2):
  - Research Site, Jena
  - Research Site, Wuppertal
- Research Site, Athens, Greece
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Nagykanizsa
  - Research Site, Nyíregyháza
  - Research Site, Zalaegerszeg
- Israel (3):
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Safed
- Japan (11):
  - Research Site, Fukuoka
  - Research Site, Koshigaya-shi
  - Research Site, Kyoto
  - Research Site, Nagoya
  - Research Site, Nara
  - Research Site, Ōita
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Tokushima
  - Research Site, Ueda-shi
  - Research Site, Utsunomiya
- Research Site, Guadalajara, Jalisco, Mexico
- Poland (3):
  - Research Site, Inowrocław
  - Research Site, Krakow
  - Research Site, Warsaw
- Research Site, Lisbon, Portugal
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
- Russia (9):
  - Research Site, Arkhangelsk
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Vsevolozhsk
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Kragujevac
- Slovakia (4):
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Trnava
  - Research Site, Žilina
- South Korea (3):
  - Research Site, Busan
  - Research Site, Seoul
  - Research Site, Wŏnju
- Taiwan (2):
  - Research Site, Chiayi City
  - Research Site, Taipei
- Research Site, Diyarbakır, Turkey (Türkiye)
- Ukraine (9):
  - Research Site, Cherkasy
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Mykolaiv
  - Research Site, Odesa
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Cheng K, Newell P, Chow JW, Broadhurst H, Wilson D, Yates K, Wardman A. Safety Profile of Ceftazidime-Avibactam: Pooled Data from the Adult Phase II and Phase III Clinical Trial Programme. Drug Saf. 2020 Aug;43(8):751-766. doi: 10.1007/s40264-020-00934-3. PMID 32602065
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- [Derived] Nichols WW, Stone GG, Newell P, Broadhurst H, Wardman A, MacPherson M, Yates K, Riccobene T, Critchley IA, Das S. Ceftazidime-Avibactam Susceptibility Breakpoints against Enterobacteriaceae and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e02590-17. doi: 10.1128/AAC.02590-17. Print 2018 Nov. PMID 30061279
- [Derived] Stone GG, Newell P, Gasink LB, Broadhurst H, Wardman A, Yates K, Chen Z, Song J, Chow JW. Clinical activity of ceftazidime/avibactam against MDR Enterobacteriaceae and Pseudomonas aeruginosa: pooled data from the ceftazidime/avibactam Phase III clinical trial programme. J Antimicrob Chemother. 2018 Sep 1;73(9):2519-2523. doi: 10.1093/jac/dky204. PMID 29912399
- [Derived] Wagenlehner FM, Sobel JD, Newell P, Armstrong J, Huang X, Stone GG, Yates K, Gasink LB. Ceftazidime-avibactam Versus Doripenem for the Treatment of Complicated Urinary Tract Infections, Including Acute Pyelonephritis: RECAPTURE, a Phase 3 Randomized Trial Program. Clin Infect Dis. 2016 Sep 15;63(6):754-762. doi: 10.1093/cid/ciw378. Epub 2016 Jun 16. PMID 27313268

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented in these forms represent the combined data base of the two identical protocols D4280C00002 and D4280C00004. The protocol D4280C00002 has a total of 522 randomized patients and the protocol D4280C00004 has a total of 511 randomized patients which adds up to a combined total of 1033 patients.
Groups:
- CAZ-AVI: Ceftazidime-avibactam treatment group
- Doripenem: Doripenem treatment group
Period: Overall Study
Arm/Group | CAZ-AVI | Doripenem
Started | 516 | 517
Completed | 473 | 476
Not Completed | 43 | 41
Not completed — Lost to Follow-up | 20 | 20
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Other Eligibility criteria | 11 | 9

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | CAZ-AVI | Doripenem | Total
Number analyzed (Participants) | 511 | 509 | 1020
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (19.76) [18 to 89] | 52.3 (18.83) [18 to 86] | 52.0 (19.29) [18 to 89]
Age, Customized [Number; unit: Participants]
  18-45 | 192 | 172 | 364
  46-64 | 162 | 177 | 339
  65-74 | 79 | 98 | 177
  75-90 | 78 | 62 | 140
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349 | 357 | 706
  Male | 162 | 152 | 314
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian Or Alaska Native | 1 | 3 | 4
  Asian | 48 | 37 | 85
  Black Or African American | 1 | 8 | 9
  Other | 40 | 35 | 75
  White | 421 | 426 | 847

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Symptomatic Response at Day 5 (mMITT Analysis Set): Non-inferiority Hypothesis Test
Description: Number of patients with symptomatic resolution (or return to premorbid state) of UTI-specific symptoms except flank pain (frequency/urgency/dysuria/suprapubic pain) with resolution of or improvement in flank pain based on the patient-reported symptom assessment response at the Day 5 visit in the mMITT analysis set. The sponsor will conclude noninferiority if the lower limit of the 95% CI of difference (corresponding to a 97.5% 1-sided lower bound) is greater than -12.5% for both FDA coprimary outcome variables (symptomatic resolution at day 5 or favorable combined response at test of cure (TOC)).
Time Frame: At Day 5 visit. Day 5 visit is based on 24 hour periods from the first dose date and time.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Symptomatic resolution | 276 | 276
  Symptom persistence | 103 | 124
  Indeterminate | 14 | 17
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: Difference (CAZ-AVI treatment group minus Doripenem treatment group) of symptomatic resolution rates ≤ non-inferiority margin; Test type: Non-Inferiority or Equivalence — -12.5%; Unstratified Miettinen & Nurminen method; Difference of symp resolution rates = 4.0, 95% CI 2-sided [-2.39 to 10.42]

2. Primary Outcome: Combined Patient-reported Symptomatic and Microbiological Response at TOC (mMITT Analysis Set): Non-inferiority Hypothesis Test
Description: Number of patients with both a favorable per patient microbiological response and symptomatic resolution (or return to premorbid state) of all UTI-specific symptoms (frequency/urgency/dysuria/suprapubic pain/flank pain) based on the patient-reported symptom assessment response at the TOC visit in the mMITT analysis set. The sponsor will conclude noninferiority if the lower limit of the 95% CI of difference (corresponding to a 97.5% 1-sided lower bound) is greater than -12.5% for both FDA coprimary outcome variables (symptomatic resolution at day 5 or favorable combined response at test of cure (TOC)).
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Favorable | 280 | 269
  Unfavorable | 81 | 109
  Indeterminate | 32 | 39
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: Difference (CAZ-AVI treatment group minus Doripenem treatment group) of favorable combined response rates ≤ non-inferiority margin; Test type: Non-Inferiority or Equivalence — -12.5%; Unstratified Miettinen & Nurminen method; Diff of favorable combined resp rates = 6.7, 95% CI 2-sided [0.30 to 13.12]

3. Primary Outcome: Per-patient Microbiological Response at TOC (mMITT Analysis Set): Non-inferiority Hypothesis Test
Description: Number of patients with a favorable per patient microbiological response at TOC. The primary efficacy outcome variable for ROW is the proportion of patients with a favorable per-patient microbiological response at the TOC visit in the mMITT analysis set.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Favorable | 304 | 296
  Unfavorable | 58 | 83
  Indeterminate | 31 | 38
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: Difference (CAZ-AVI treatment group minus Doripenem treatment group) of favorable response rates ≤ non-inferiority margin; Test type: Non-Inferiority or Equivalence — -12.5%; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 6.4, 95% CI 2-sided [0.33 to 12.36]

4. Secondary Outcome: Per-patient Microbiological Response at EOT (IV) (mMITT Analysis Set)
Description: Number of patients with a favorable per-patient microbiological response at EOT (IV)
Time Frame: At EOT (IV) visit. EOT (IV) visit is Within 24 hours after completion of the last infusion of IV study therapy and on/before the first dose for oral study therapy
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Favorable | 374 | 395
  Unfavorable | 1 | 3
  Indeterminate | 18 | 19
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of favorable response rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 0.4, 95% CI 2-sided [-2.70 to 3.56]

5. Secondary Outcome: Per-patient Microbiological Response at LFU (mMITT Analysis Set)
Description: Number of patients with a favorable per patient microbiological response at LFU
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Favorable | 268 | 254
  Unfavorable | 83 | 125
  Indeterminate | 42 | 38
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 7.3, 95% CI 2-sided [0.68 to 13.81]

6. Secondary Outcome: Per-patient Microbiological Response at EOT (IV) (ME at EOT (IV) Analysis Set)
Description: Number of patients with a favorable per-patient microbiological response at EOT (IV)
Time Frame: as for outcome 4
Population: Microbiological evaluable analysis set at EOT (IV) (ME at EOT (IV))
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 325 | 361
Participants
  Favorable | 324 | 359
  Unfavorable | 1 | 2
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 0.2, 95% CI 2-sided [-1.21 to 1.72]

7. Secondary Outcome: Per-patient Microbiological Response at TOC (ME at TOC Analysis Set)
Description: Number of patients with a favorable per patient microbiological response at TOC
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological evaluable analysis set at TOC (ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participants
  Favorable | 241 | 225
  Unfavorable | 45 | 73
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 8.8, 95% CI 2-sided [2.27 to 15.24]

8. Secondary Outcome: Per-patient Microbiological Response at LFU (ME at LFU Analysis Set)
Description: Number of patients with a favorable per patient microbiological response at LFU
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Microbiological evaluable analysis set at LFU (ME at LFU)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 245 | 262
Participants
  Favorable | 182 | 166
  Unfavorable | 63 | 96
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 10.9, 95% CI 2-sided [2.86 to 18.85]

9. Secondary Outcome: Per-patient Microbiological Response at EOT (IV) (Extended ME at EOT (IV) Analysis Set)
Description: Number of patients with a favorable per-patient microbiological response at EOT (IV)
Time Frame: as for outcome 4
Population: Extended microbiological evaluable analysis set at EOT (IV) (EME at EOT (IV))
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 336 | 371
Participants
  Favorable | 335 | 369
  Unfavorable | 1 | 2
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 0.2, 95% CI 2-sided [-1.17 to 1.68]

10. Secondary Outcome: Per-patient Microbiological Response at TOC (Extended ME at TOC Analysis Set)
Description: Number of patients with a favorable per patient microbiological response at TOC
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Extended microbiological evaluable analysis set at TOC (Extended ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participants
  Favorable | 243 | 236
  Unfavorable | 49 | 75
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 7.3, 95% CI 2-sided [0.88 to 13.74]

11. Secondary Outcome: Per-patient Microbiological Response at LFU (Extended ME at LFU Analysis Set)
Description: Number of patients with a favorable per patient microbiological response at LFU
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Extended microbiological evaluable analysis set at LFU (Extended ME at LFU)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 251 | 272
Participants
  Favorable | 184 | 173
  Unfavorable | 67 | 99
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 9.7, 95% CI 2-sided [1.72 to 17.55]

12. Secondary Outcome: Investigator Determined Clinical Response at EOT (IV) (mMITT Analysis Set)
Description: Number of patients with a clinical cure at EOT (IV). The investigator should consider the entirety of the patient's clinical course and current status, including an evaluation of signs and symptoms (eg, fever, dysuria, costovertebral angle tenderness) and physical examination in order to classify the patient's clinical response.
Time Frame: as for outcome 4
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Clinical cure | 378 | 407
  Clinical failure | 5 | 5
  Indeterminate | 10 | 5
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = -1.4, 95% CI 2-sided [-4.07 to 1.02]

13. Secondary Outcome: Investigator Determined Clinical Response at TOC (mMITT Analysis Set)
Description: Number of patients with a clinical cure at TOC. The investigator should consider the entirety of the patient's clinical course and current status, including an evaluation of signs and symptoms (eg, fever, dysuria, costovertebral angle tenderness) and physical examination in order to classify the patient's clinical response.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Clinical cure | 355 | 377
  Clinical failure | 11 | 24
  Indeterminate | 27 | 16
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = -0.1, 95% CI 2-sided [-4.23 to 4.03]

14. Secondary Outcome: Investigator Determined Clinical Response at LFU (mMITT Analysis Set)
Description: Number of patients with a clinical cure at LFU. The investigator should consider the entirety of the patient's clinical course and current status, including an evaluation of signs and symptoms (eg, fever, dysuria, costovertebral angle tenderness) and physical examination in order to classify the patient's clinical response.
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Clinical cure | 335 | 350
  Clinical failure | 23 | 39
  Indeterminate | 35 | 28
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 1.3, 95% CI 2-sided [-3.71 to 6.30]

15. Secondary Outcome: Investigator Determined Clinical Response at EOT (IV) (ME at EOT (IV) Analysis Set)
Description: as for outcome 12
Time Frame: as for outcome 4
Population: Microbiological evaluable analysis set at EOT (IV) (ME at EOT (IV))
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 325 | 361
Participants
  Clinical cure | 318 | 358
  Clinical failure | 4 | 2
  Indeterminate | 3 | 1
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = -1.3, 95% CI 2-sided [-3.64 to 0.55]

16. Secondary Outcome: Investigator Determined Clinical Response at TOC (ME at TOC Analysis Set)
Description: as for outcome 13
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological evaluable analysis set at TOC (ME at TOC )
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participants
  Clinical cure | 277 | 285
  Clinical failure | 4 | 13
  Indeterminate | 5 | 0
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 1.2, 95% CI 2-sided [-2.03 to 4.56]

17. Secondary Outcome: Investigator Determined Clinical Response at LFU (ME at LFU Analysis Set)
Description: as for outcome 14
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Microbiological evaluable analysis set at LFU (ME at LFU)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 245 | 262
Participants
  Clinical cure | 226 | 236
  Clinical failure | 15 | 24
  Indeterminate | 4 | 2
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 2.2, 95% CI 2-sided [-2.90 to 7.24]

18. Secondary Outcome: Investigator Determined Clinical Response at EOT (IV) (Extended ME at EOT (IV) Analysis Set)
Description: as for outcome 12
Time Frame: as for outcome 4
Population: Extended microbiological evaluable analysis set at EOT (IV) (Extended ME at EOT (IV))
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 336 | 371
Participants
  Clinical cure | 327 | 368
  Clinical failure | 4 | 2
  Indeterminate | 5 | 1
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = -1.9, 95% CI 2-sided [-4.30 to 0.04]

19. Secondary Outcome: Investigator Determined Clinical Response at TOC (Extended ME at TOC Analysis Set)
Description: as for outcome 13
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Extended microbiological evaluable analysis set at TOC (Extended ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participants
  Clinical cure | 283 | 298
  Clinical failure | 4 | 13
  Indeterminate | 5 | 0
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 1.1, 95% CI 2-sided [-2.07 to 4.32]

20. Secondary Outcome: Investigator Determined Clinical Response at LFU (Extended ME at LFU Analysis Set)
Description: as for outcome 14
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Extended microbiological evaluable analysis set at LFU (Extended ME at LFU)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 251 | 272
Participants
  Clinical cure | 232 | 246
  Clinical failure | 15 | 24
  Indeterminate | 4 | 2
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 2.0, 95% CI 2-sided [-2.94 to 6.91]

21. Secondary Outcome: Investigator Determined Clinical Response at EOT (IV) (CE at EOT (IV) Analysis Set)
Description: as for outcome 12
Time Frame: as for outcome 4
Population: Clinically evaluable analysis set at EOT (IV) (CE at EOT (IV))
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 350 | 391
Participants
  Clinical cure | 346 | 387
  Clinical failure | 4 | 4
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = -0.1, 95% CI 2-sided [-1.99 to 1.61]

22. Secondary Outcome: Investigator Determined Clinical Response at TOC (CE at TOC Analysis Set)
Description: as for outcome 13
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Clinically evaluable analysis set at TOC (CE at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 297 | 330
Participants
  Clinical cure | 289 | 309
  Clinical failure | 8 | 21
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 3.7, 95% CI 2-sided [0.41 to 7.16]

23. Secondary Outcome: Investigator Determined Clinical Response at LFU (CE at LFU Analysis Set)
Description: as for outcome 14
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Clinically evaluable analysis set at LFU (CE at LFU)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 254 | 287
Participants
  Clinical cure | 235 | 254
  Clinical failure | 19 | 33
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clinical cure rates = 4.0, 95% CI 2-sided [-1.00 to 9.05]

24. Secondary Outcome: Investigator Determined Clinical Response at TOC for Patients Infected by Ceftazidime-resistant Gram-negative Pathogen (mMITT Analysis Set)
Description: Clinical cure at the TOC visit for patients infected with a ceftazidime resistant pathogen in the mMITT analysis set. Includes patients infected by at least one ceftazidime-resistant Gram-negative pathogen.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  All patients - Clinical cure (n=75, 84) | 67 | 75
  Escherichia coli patients - Clin cure (n=36, 37) | 33 | 31
  Klebsiella pneumoniae patients-Clin cure(n=18,30) | 17 | 28
  Pseudomonas aeruginosa patients- Clin cure(n=7,6) | 5 | 6
  Enterobacter cloacae patients-Clin cure(n=7,6) | 5 | 5
  Proteus mirabilis patients - Clin cure (n=2, 5) | 2 | 5
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; Confidence interval of the difference (CAZ-AVI treatment group minus Doripenem treatment group) of clinical cure rates in All patients with a ceftazidime-resistant Gram-negative pathogen; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clin cure rates in All patients = 0.0, 95% CI 2-sided [-10.4 to 10.1]

25. Secondary Outcome: Investigator Determined Clinical Response at TOC for Patients Infected by Ceftazidime-resistant Gram-negative Pathogen (ME at TOC Analysis Set)
Description: Clinical cure at the TOC visit for patients infected with a ceftazidime resistant pathogen in the ME at TOC analysis set. Includes patients infected by at least one ceftazidime-resistant Gram-negative pathogen.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological evaluable analysis set at TOC(ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participants
  All patients - Clinical cure (n=48, 57) | 47 | 55
  Escherichia coli patients-Clin cure (n=23,27) | 22 | 25
  Klebsiella pneumoniae patients-Clin cure(n=14, 22) | 14 | 22
  Pseudomonas aeruginosa patients-Clin cure(n=1, 2) | 1 | 2
  Enterobacter cloacae patients-Clin cure(n=5,5) | 5 | 5
  Proteus mirabilis patients - Clin cure (n=0, 2) | 0 | 2
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clin cure rates in All patients = 1.4, 95% CI 2-sided [-7.8 to 10.2]

26. Secondary Outcome: Investigator Determined Clinical Response at TOC for Patients Infected by Ceftazidime-resistant Gram-negative Pathogen (Extended ME at TOC Analysis Set)
Description: Clinical cure at the TOC visit for patients infected with a ceftazidime resistant pathogen in the Extended ME at TOC analysis set. Includes patients infected by at least one ceftazidime-resistant Gram-negative pathogen.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Extended microbiological evaluable analysis set at TOC(Extended ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participants
  All patients - Clinical cure (n=51, 63) | 50 | 61
  Escherichia coli patients - Clin cure (n=23, 27) | 22 | 25
  Klebsiella pneumoniae patients-Clin cure(n=15, 23) | 15 | 23
  Pseudomonas aeruginosa patients-Clin cure(n=3,6) | 3 | 6
  Enterobacter cloacae patients-Clin cure(n=5,5) | 5 | 5
  Proteus mirabilis patients - Clin cure (n=0, 2) | 0 | 2
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of clin cure rates in All patients = 1.2, 95% CI 2-sided [-7.5 to 9.2]

27. Secondary Outcome: Per-patient Microbiological Response at TOC in Patients Infected by Ceftazidime-resistant Gram-negative Pathogen (mMITT Analysis Set)
Description: Favorable per-patient microbiological response at the TOC visit for patients infected with a ceftazidime resistant pathogen in the mMITT analysis set.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 75 | 84
Participants
  Favorable | 47 | 51
  Unfavorable | 19 | 27
  Indeterminate | 9 | 6
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 2.0, 95% CI 2-sided [-13.18 to 16.89]

28. Secondary Outcome: Per-patient Microbiological Response at TOC in Patients Infected by Ceftazidime-resistant Gram-negative Pathogen (ME at TOC Analysis Set)
Description: Favorable per-patient microbiological response at the TOC visit for patients infected with a ceftazidime resistant pathogen in the ME at TOC analysis set.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological evaluable analysis set at TOC(ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 48 | 57
Participants
  Favorable | 35 | 37
  Unfavorable | 13 | 20
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 8.0, 95% CI 2-sided [-10.03 to 25.21]

29. Secondary Outcome: Per-patient Microbiological Response at TOC in Patients Infected by Ceftazidime-resistant Gram-negative Pathogen (Extended ME at TOC Analysis Set)
Description: Favorable per-patient microbiological response at the TOC visit for patients infected with a ceftazidime resistant pathogen in the Extended ME at TOC analysis set.
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Extended microbiological evaluable analysis set at TOC(Extended ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 51 | 63
Participants
  Favorable | 37 | 41
  Unfavorable | 14 | 22
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Unstratified Miettinen & Nurminen method; Diff of favorable response rates = 7.5, 95% CI 2-sided [-9.91 to 24.01]

30. Secondary Outcome: Time to First Defervescence While on IV Study Therapy (mMITT Analysis Set)
Description: Time to first defervescence while on IV study therapy in patients in the mMITT analysis set who have fever at study entry.
Time Frame: Time to first defervescence is defined as the time (in days) from the first dose of IV study therapy to first absence of fever, which is temperature ≤ 37.8 C in a 24-hour period.
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participants
  Number of patients with fever (>38°C) at baseline | 157 | 150
  Number afebrile at the time of the last obs | 155 | 143
  Number censored at the time of the last obs | 2 | 7
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: No difference in time to first defervescence between treatment groups; Test type: Superiority or Other; p = 0.038, Log Rank

31. Secondary Outcome: Time to First Defervescence While on IV Study Therapy (ME at TOC Analysis Set)
Description: Time to first defervescence while on IV study therapy in patients in the ME at TOC analysis set who have fever at study entry.
Time Frame: as for outcome 30
Population: Microbiological evaluable analysis set at TOC(ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participants
  Number of patients with fever (>38°C) at baseline | 124 | 108
  Number afebrile at the time of the last obs | 124 | 105
  Number censored at the time of the last obs | 0 | 3
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: No difference in time to first defervescence between treatment groups; Test type: Superiority or Other; p = 0.129, Log Rank

32. Secondary Outcome: Time to First Defervescence While on IV Study Therapy (Extended ME at TOC Analysis Set)
Description: Time to first defervescence while on IV study therapy in patients in the Extended ME at TOC analysis set who have fever at study entry.
Time Frame: as for outcome 30
Population: Extended microbiological evaluable analysis set at TOC(Extended ME at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participants
  Number of patients with fever (>38°C) at baseline | 124 | 111
  Number afebrile at the time of the last obs | 124 | 108
  Number censored at the time of the last obs | 0 | 3
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: No difference in time to first defervescence between treatment groups; Test type: Superiority or Other; p = 0.080, Log Rank

33. Secondary Outcome: Time to First Defervescence While on IV Study Therapy (CE at TOC Analysis Set)
Description: Time to first defervescence while on IV study therapy in patients in the CE at TOC analysis set who have fever at study entry.
Time Frame: as for outcome 30
Population: Clinically evaluable analysis set at TOC(CE at TOC)
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 297 | 330
Participants
  Number of patients with fever (>38°C) at baseline | 123 | 118
  Number afebrile at the time of the last obs | 122 | 113
  Number censored at the time of the last obs | 1 | 5
Statistical Analysis 1: Comparison: CAZ-AVI vs Doripenem; H0: No difference in time to first defervescence between treatment groups; Test type: Superiority or Other; p = 0.155, Log Rank

34. Secondary Outcome: Per-pathogen Microbiological Response at EOT (IV) for Baseline Pathogen (mMITT Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the EOT (IV) visit in the mMITT analysis set
Time Frame: At EOT IV visit. EOT (IV) visit is Within 24 hours after completion of the last infusion of IV study therapy and on/before the first dose for oral study therapy
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  Escherichia coli - Favorable (n=292, 306) | 280 | 293
  Klebsiella pneumoniae - Favorable (n=44, 56) | 41 | 51
  Proteus mirabilis - Favorable (n=17, 13) | 16 | 11
  Enterobacter cloacae - Favorable (n= 11,13) | 9 | 13
  Pseudomonas aeruginosa - Favorable (n=18, 20) | 17 | 18

35. Secondary Outcome: Per-pathogen Microbiological Response at TOC for Baseline Pathogen (mMITT Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the TOC visit in the mMITT analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  Escherichia coli - Favorable (n=292, 306) | 229 | 220
  Klebsiella pneumoniae - Favorable (n=44, 56) | 33 | 35
  Proteus mirabilis - Favorable (n=17, 13) | 16 | 9
  Enterobacter cloacae - Favorable (n= 11,13) | 6 | 9
  Pseudomonas aeruginosa - Favorable (n=18, 20) | 12 | 15

36. Secondary Outcome: Per-pathogen Microbiological Response at LFU for Baseline Pathogen (mMITT Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the LFU visit in the mMITT analysis set
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  Escherichia coli - Favorable (n=292, 306) | 198 | 189
  Klebsiella pneumoniae - Favorable (n=44, 56) | 32 | 30
  Proteus mirabilis - Favorable (n=17, 13) | 16 | 6
  Enterobacter cloacae - Favorable (n= 11,13) | 6 | 9
  Pseudomonas aeruginosa - Favorable (n=18, 20) | 9 | 13

37. Secondary Outcome: Per-pathogen Microbiological Response at EOT (IV) for Baseline Pathogen (Extended ME at EOT (IV) Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the EOT (IV) visit in the Extended ME at EOT (IV) analysis set
Time Frame: as for outcome 34
Population: Extended microbiological evaluable analysis set at EOT (IV) (EME at EOT (IV))
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 336 | 371
Participant
  Escherichia coli - Favorable (n=250, 274) | 250 | 274
  Klebsiella pneumoniae - Favorable (n=34, 49) | 34 | 48
  Proteus mirabilis - Favorable (n=13, 11) | 13 | 11
  Enterobacter cloacae - Favorable (n= 9, 12) | 9 | 12
  Pseudomonas aeruginosa - Favorable (n=18, 18) | 17 | 17

38. Secondary Outcome: Per-pathogen Microbiological Response at TOC for Baseline Pathogen (Extended ME at TOC Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the TOC visit in the Extended ME at TOC analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Extended microbiological evaluable analysis set at TOC (EME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participant
  Escherichia coli - Favorable (n=214, 226) | 180 | 176
  Klebsiella pneumoniae - Favorable (n=32, 42) | 26 | 29
  Proteus mirabilis - Favorable (n=14, 7) | 14 | 4
  Enterobacter cloacae - Favorable (n= 7, 11) | 5 | 8
  Pseudomonas aeruginosa - Favorable (n=13, 18) | 8 | 13

39. Secondary Outcome: Per-pathogen Microbiological Response at LFU for Baseline Pathogen (Extended ME at LFU Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the LFU visit in the Extended ME at LFU analysis set
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Extended microbiological evaluable analysis set at LFU (EME at LFU)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 251 | 272
Participant
  Escherichia coli - Favorable (n=179, 198) | 129 | 131
  Klebsiella pneumoniae - Favorable (n=31, 36) | 24 | 19
  Proteus mirabilis - Favorable (n=11,5) | 11 | 1
  Enterobacter cloacae - Favorable (n= 7, 11) | 5 | 8
  Pseudomonas aeruginosa - Favorable (n=12, 16) | 7 | 9

40. Secondary Outcome: Per-pathogen Microbiological Response at EOT (IV) for Baseline Pathogen (ME at EOT (IV) Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the EOT (IV) visit in the ME at EOT (IV) analysis set
Time Frame: as for outcome 4
Population: Microbiological evaluable analysis set at EOT (IV) (ME at EOT (IV))
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 325 | 361
Participant
  Escherichia coli - Favorable (n=249, 270) | 249 | 270
  Klebsiella pneumoniae - Favorable (n=33, 48) | 33 | 47
  Proteus mirabilis - Favorable (n=13,11) | 13 | 11
  Enterobacter cloacae - Favorable (n= 9, 12) | 9 | 12
  Pseudomonas aeruginosa - Favorable (n=10, 15) | 9 | 14

41. Secondary Outcome: Per-pathogen Microbiological Response at TOC for Baseline Pathogen (ME at TOC Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the TOC visit in the ME at TOC analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological evaluable analysis set at TOC (ME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participant
  Escherichia coli - Favorable (n=214, 221) | 180 | 171
  Klebsiella pneumoniae - Favorable (n=31, 41) | 25 | 28
  Proteus mirabilis - Favorable (n=14, 7) | 14 | 4
  Enterobacter cloacae - Favorable (n= 7, 11) | 5 | 8
  Pseudomonas aeruginosa - Favorable (n=9, 13) | 7 | 9

42. Secondary Outcome: Per-pathogen Microbiological Response at LFU for Baseline Pathogen (ME at LFU Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the LFU visit in the ME at LFU analysis set
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Microbiological evaluable analysis set at LFU (ME at LFU)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 245 | 262
Participant
  Escherichia coli - Favorable (n=179, 194) | 129 | 127
  Klebsiella pneumoniae - Favorable (n=30, 35) | 23 | 18
  Proteus mirabilis - Favorable (n=11,5) | 11 | 1
  Enterobacter cloacae - Favorable (n= 7, 11) | 5 | 8
  Pseudomonas aeruginosa - Favorable (n=8, 13) | 6 | 8

43. Secondary Outcome: Per-pathogen Microbiological Response at EOT (IV) for Blood Only (mMITT Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the EOT (IV) visit in the mMITT analysis set for blood only
Time Frame: as for outcome 34
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  Escherichia coli - Favorable (n=32, 28) | 31 | 28
  Klebsiella pneumoniae - Favorable (n=4, 2) | 2 | 2
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=1, 2) | 1 | 2

44. Secondary Outcome: Per-pathogen Microbiological Response at TOC for Blood Only (mMITT Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the TOC visit in the mMITT analysis set for blood only
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  Escherichia coli - Favorable (n=32, 28) | 31 | 28
  Klebsiella pneumoniae - Favorable (n=4, 2) | 3 | 2
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=1, 2) | 1 | 2

45. Secondary Outcome: Per-pathogen Microbiological Response at LFU for Blood Only (mMITT Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the LFU visit in the mMITT analysis set for blood only
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  Escherichia coli - Favorable (n=32, 28) | 29 | 27
  Klebsiella pneumoniae - Favorable (n=4, 2) | 3 | 2
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=1, 2) | 1 | 2

46. Secondary Outcome: Per-pathogen Microbiological Response at EOT (IV) for Blood Only (Extended ME at EOT (IV) Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the EOT (IV) visit in the Extended ME at EOT (IV) analysis set for blood only
Time Frame: as for outcome 34
Population: Extended microbiological evaluable analysis set at EOT (IV) (EME at EOT (IV))
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 336 | 371
Participant
  Escherichia coli - Favorable (n=26, 24) | 26 | 24
  Klebsiella pneumoniae - Favorable (n=2, 1) | 1 | 1
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=1, 2) | 1 | 2

47. Secondary Outcome: Per-pathogen Microbiological Response at TOC for Blood Only (Extended ME at TOC Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the TOC visit in the Extended ME at TOC analysis set for blood only
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Extended microbiological evaluable analysis set at TOC (EME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participant
  Escherichia coli - Favorable (n=22, 20) | 22 | 20
  Klebsiella pneumoniae - Favorable (n=2, 2) | 2 | 2
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=0, 1) | 0 | 1

48. Secondary Outcome: Per-pathogen Microbiological Response at LFU for Blood Only (Extended ME at LFU Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the LFU visit in the Extended ME at LFU analysis set for blood only
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Extended microbiological evaluable analysis set at LFU (EME at LFU)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 251 | 272
Participant
  Escherichia coli - Favorable (n=19, 18) | 19 | 17
  Klebsiella pneumoniae - Favorable (n=2, 1) | 2 | 1
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=0, 1) | 0 | 1

49. Secondary Outcome: Per-pathogen Microbiological Response at EOT (IV) for Blood Only (ME at EOT (IV) Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the EOT (IV) visit in the ME at EOT (IV) analysis set for blood only
Time Frame: as for outcome 4
Population: Microbiological evaluable analysis set at EOT (IV) (ME at EOT (IV))
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 325 | 361
Participant
  Escherichia coli - Favorable (n=26, 24) | 26 | 24
  Klebsiella pneumoniae - Favorable (n=2, 1) | 1 | 1
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=1, 2) | 1 | 2

50. Secondary Outcome: Per-pathogen Microbiological Response at TOC for Blood Only (ME at TOC Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the TOC visit in the ME at TOC analysis set for blood only
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization.
Population: Microbiological evaluable analysis set at TOC (ME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participant
  Escherichia coli - Favorable (n=22, 20) | 22 | 20
  Klebsiella pneumoniae - Favorable (n=2, 2) | 2 | 2
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=0, 1) | 0 | 1

51. Secondary Outcome: Per-pathogen Microbiological Response at LFU for Blood Only (ME at LFU Analysis Set)
Description: Number of favorable per-pathogen microbiological responses at the LFU visit in the ME at LFU analysis set for blood only
Time Frame: At LFU visit. LFU visit is 45 to 52 days from Randomization.
Population: Microbiological evaluable analysis set at LFU (ME at LFU)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 245 | 262
Participant
  Escherichia coli - Favorable (n=19, 18) | 19 | 17
  Klebsiella pneumoniae - Favorable (n=2, 1) | 2 | 1
  Proteus mirabilis - Favorable (n=1, 0) | 1 | 0
  Pseudomonas aeruginosa - Favorable (n=0, 1) | 0 | 1

52. Secondary Outcome: Per-pathogen Microbiological Response at TOC by CAZ AVI MIC for Baseline Pathogen (mMITT Analysis Set)
Description: Per pathogen microbiological response at TOC by CAZ-AVI MIC for baseline pathogen in the mMITT analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  E. coli (MIC: <=0.008) - Favorable (n=5, 6) | 3 | 5
  E. coli (MIC: 0.015) - Favorable (n=8, 7) | 8 | 6
  E. coli (MIC: 0.03) - Favorable (n=28, 35) | 24 | 23
  E. coli (MIC: 0.06) - Favorable (n=123, 139) | 103 | 111
  E. coli (MIC: 0.12) - Favorable (n=90, 81) | 67 | 54
  E. coli (MIC: 0.25) - Favorable (n=28, 25) | 18 | 13
  E. coli (MIC: 0.5) - Favorable (n=5, 6) | 4 | 2
  E. coli (MIC: 1) - Favorable (n=3, 0) | 1 | 0
  E. coli (MIC: 2) - Favorable (n=1, 0) | 1 | 0
  E. coli (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 32) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: >32) - Favorable (n=0, 0) | 0 | 0
  Kleb.pneumoniae (MIC: <=0.008)-Favorable(n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 0.015) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 0.03) - Favorable (n=1, 2) | 1 | 2
  Kleb. pneumoniae (MIC: 0.06) - Favorable (n=9, 8) | 7 | 8
  Kleb.pneumoniae (MIC: 0.12) -Favorable(n=11, 10) | 9 | 7
  Kleb. pneumoniae (MIC: 0.25) - Favorable (n=4, 10) | 1 | 3
  Kleb. pneumoniae (MIC: 0.5) - Favorable (n=8, 16) | 6 | 11
  Kleb. pneumoniae (MIC: 1) - Favorable (n=8, 5) | 6 | 3
  Kleb. pneumoniae (MIC: 2) - Favorable (n= 2, 4) | 2 | 0
  Kleb. pneumoniae (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 32) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: >32) - Favorable (n=0, 1) | 0 | 1
  Proteus mirabilis (MIC:<=0.008)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.015)- Favorable (n=1,1) | 1 | 0
  Proteus mirabilis (MIC: 0.03)- Favorable (n=10, 5) | 10 | 3
  Proteus mirabilis (MIC: 0.06)- Favorable (n=6,6) | 5 | 5
  Proteus mirabilis (MIC: 0.12)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.25)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 0.5)- Favorable (n=0,1) | 0 | 1
  Proteus mirabilis (MIC: 1)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 2)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 4)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 8)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 16)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 32)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: >32)- Favorable (n=0, 0) | 0 | 0
  Entero. cloacae (MIC: <=0.008)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.015)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.03)- Favorable (n= 1,0) | 1 | 0
  Entero. cloacae (MIC: 0.06)- Favorable (n= 0, 1) | 0 | 1
  Entero. cloacae (MIC: 0.12)- Favorable (n= 3,2) | 2 | 2
  Entero. cloacae (MIC: 0.25)- Favorable (n= 1,4) | 0 | 1
  Entero. cloacae (MIC: 0.5)- Favorable (n= 1,1) | 0 | 1
  Entero. cloacae (MIC: 1)- Favorable (n= 2,5) | 1 | 4
  Entero. cloacae (MIC: 2)- Favorable (n= 1,0) | 1 | 0
  Entero. cloacae (MIC: 4)- Favorable (n= 2,0) | 1 | 0
  Entero. cloacae (MIC: 8)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 16)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 32)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: >32)- Favorable (n= 0,0) | 0 | 0
  P.aeruginosa (MIC: <=0.008) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.015) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.03) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.06) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.12) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.25) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.5) - Favorable (n=0,2) | 0 | 2
  P.aeruginosa (MIC: 1) - Favorable (n=1,4) | 1 | 2
  P.aeruginosa (MIC: 2) - Favorable (n=5,5) | 5 | 5
  P.aeruginosa (MIC: 4) - Favorable (n=7,6) | 3 | 4
  P.aeruginosa (MIC: 8) - Favorable (n=2,2) | 1 | 1
  P.aeruginosa (MIC: 16) - Favorable (n=1,1) | 0 | 1
  P.aeruginosa (MIC: 32) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: >32) - Favorable (n=2,0) | 2 | 0

53. Secondary Outcome: Per-pathogen Microbiological Response at TOC by CAZ AVI MIC for Baseline Pathogen (Extended ME at TOC Analysis Set)
Description: Per pathogen microbiological response at TOC by CAZ-AVI MIC for baseline pathogen in the Extended ME at TOC analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Extended microbiological evaluable analysis set at TOC (EME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participant
  E. coli (MIC: <=0.008) - Favorable (n=4,4) | 2 | 4
  E. coli (MIC: 0.015) - Favorable (n=5, 6) | 5 | 5
  E. coli (MIC: 0.03) - Favorable (n=18, 21) | 17 | 17
  E. coli (MIC: 0.06) - Favorable (n=95, 111) | 83 | 94
  E. coli (MIC: 0.12) - Favorable (n=68, 54) | 56 | 40
  E. coli (MIC: 0.25) - Favorable (n=19, 18) | 13 | 8
  E. coli (MIC: 0.5) - Favorable (n=2, 5) | 2 | 2
  E. coli (MIC: 1) - Favorable (n=2, 0) | 1 | 0
  E. coli (MIC: 2) - Favorable (n=1, 0) | 1 | 0
  E. coli (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 32) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: >32) - Favorable (n=0, 0) | 0 | 0
  Kleb.pneumoniae (MIC: <=0.008)-Favorable(n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 0.015) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 0.03) - Favorable (n=1, 2) | 1 | 2
  Kleb. pneumoniae (MIC: 0.06) - Favorable (n=5, 7) | 4 | 7
  Kleb.pneumoniae (MIC: 0.12) -Favorable(n=8, 9) | 7 | 6
  Kleb. pneumoniae (MIC: 0.25) - Favorable (n=3, 7) | 1 | 2
  Kleb. pneumoniae (MIC: 0.5) - Favorable (n=6, 11) | 4 | 8
  Kleb. pneumoniae (MIC: 1) - Favorable (n=6, 4) | 6 | 3
  Kleb. pneumoniae (MIC: 2) - Favorable (n= 2, 1) | 2 | 0
  Kleb. pneumoniae (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 32) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: >32) - Favorable (n=0, 1) | 0 | 1
  Proteus mirabilis (MIC:<=0.008)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.015)- Favorable (n=1,0) | 1 | 0
  Proteus mirabilis (MIC: 0.03)- Favorable (n=9, 2) | 9 | 0
  Proteus mirabilis (MIC: 0.06)- Favorable (n=4,5) | 4 | 4
  Proteus mirabilis (MIC: 0.12)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.25)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 0.5)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 1)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 2)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 4)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 8)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 16)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 32)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: >32)- Favorable (n=0, 0) | 0 | 0
  Entero. cloacae (MIC: <=0.008)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.015)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.03)- Favorable (n= 1,0) | 1 | 0
  Entero. cloacae (MIC: 0.06)- Favorable (n= 0, 1) | 0 | 1
  Entero. cloacae (MIC: 0.12)- Favorable (n= 1,2) | 1 | 2
  Entero. cloacae (MIC: 0.25)- Favorable (n= 0,3) | 0 | 0
  Entero. cloacae (MIC: 0.5)- Favorable (n= 1,1) | 0 | 1
  Entero. cloacae (MIC: 1)- Favorable (n= 1,4) | 1 | 4
  Entero. cloacae (MIC: 2)- Favorable (n= 1,0) | 1 | 0
  Entero. cloacae (MIC: 4)- Favorable (n= 2,0) | 1 | 0
  Entero. cloacae (MIC: 8)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 16)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 32)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: >32)- Favorable (n= 0,0) | 0 | 0
  P.aeruginosa (MIC: <=0.008) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.015) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.03) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.06) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.12) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.25) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.5) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 1) - Favorable (n=1,4) | 1 | 2
  P.aeruginosa (MIC: 2) - Favorable (n=4,5) | 4 | 5
  P.aeruginosa (MIC: 4) - Favorable (n=5,6) | 1 | 4
  P.aeruginosa (MIC: 8) - Favorable (n=2,2) | 1 | 1
  P.aeruginosa (MIC: 16) - Favorable (n=0,1) | 0 | 1
  P.aeruginosa (MIC: 32) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: >32) - Favorable (n=1,0) | 1 | 0

54. Secondary Outcome: Per-pathogen Microbiological Response at TOC by CAZ AVI MIC for Baseline Pathogen (ME at TOC Analysis Set)
Description: Per pathogen microbiological response at TOC by CAZ-AVI MIC for baseline pathogen in the ME at TOC analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Microbiological evaluable analysis set at TOC (ME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participant
  E. coli (MIC: <=0.008) - Favorable (n=4,4) | 2 | 4
  E. coli (MIC: 0.015) - Favorable (n=5, 6) | 5 | 5
  E. coli (MIC: 0.03) - Favorable (n=18, 21) | 17 | 17
  E. coli (MIC: 0.06) - Favorable (n=95, 111) | 83 | 94
  E. coli (MIC: 0.12) - Favorable (n=68, 54) | 56 | 40
  E. coli (MIC: 0.25) - Favorable (n=19, 18) | 13 | 8
  E. coli (MIC: 0.5) - Favorable (n=2, 5) | 2 | 2
  E. coli (MIC: 1) - Favorable (n=2, 0) | 1 | 0
  E. coli (MIC: 2) - Favorable (n=1, 0) | 1 | 0
  E. coli (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 32) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: >32) - Favorable (n=0, 0) | 0 | 0
  Kleb.pneumoniae (MIC: <=0.008)-Favorable(n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 0.015) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 0.03) - Favorable (n=1, 2) | 1 | 2
  Kleb. pneumoniae (MIC: 0.06) - Favorable (n=5, 7) | 4 | 7
  Kleb.pneumoniae (MIC: 0.12) -Favorable(n=8, 9) | 7 | 6
  Kleb. pneumoniae (MIC: 0.25) - Favorable (n=3, 7) | 1 | 2
  Kleb. pneumoniae (MIC: 0.5) - Favorable (n=6, 11) | 4 | 8
  Kleb. pneumoniae (MIC: 1) - Favorable (n=5, 4) | 5 | 3
  Kleb. pneumoniae (MIC: 2) - Favorable (n= 2, 1) | 2 | 0
  Kleb. pneumoniae (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 32) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: >32) - Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC:<=0.008)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.015)- Favorable (n=1,0) | 1 | 0
  Proteus mirabilis (MIC: 0.03)- Favorable (n=9, 2) | 9 | 0
  Proteus mirabilis (MIC: 0.06)- Favorable (n=4,5) | 4 | 4
  Proteus mirabilis (MIC: 0.12)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.25)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 0.5)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 1)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 2)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 4)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 8)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 16)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 32)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: >32)- Favorable (n=0, 0) | 0 | 0
  Entero. cloacae (MIC: <=0.008)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.015)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.03)- Favorable (n= 1,0) | 1 | 0
  Entero. cloacae (MIC: 0.06)- Favorable (n= 0, 1) | 0 | 1
  Entero. cloacae (MIC: 0.12)- Favorable (n= 1,2) | 1 | 2
  Entero. cloacae (MIC: 0.25)- Favorable (n= 0,3) | 0 | 0
  Entero. cloacae (MIC: 0.5)- Favorable (n= 1,1) | 0 | 1
  Entero. cloacae (MIC: 1)- Favorable (n= 1,4) | 1 | 4
  Entero. cloacae (MIC: 2)- Favorable (n= 1,0) | 1 | 0
  Entero. cloacae (MIC: 4)- Favorable (n= 2,0) | 1 | 0
  Entero. cloacae (MIC: 8)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 16)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 32)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: >32)- Favorable (n= 0,0) | 0 | 0
  P.aeruginosa (MIC: <=0.008) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.015) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.03) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.06) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.12) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.25) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.5) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 1) - Favorable (n=1,4) | 1 | 2
  P.aeruginosa (MIC: 2) - Favorable (n=4,4) | 4 | 4
  P.aeruginosa (MIC: 4) - Favorable (n=3,4) | 1 | 3
  P.aeruginosa (MIC: 8) - Favorable (n=1,1) | 1 | 0
  P.aeruginosa (MIC: 16) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 32) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: >32) - Favorable (n=0,0) | 0 | 0

55. Secondary Outcome: Per-pathogen Microbiological Response at TOC by Doripenem MIC for Baseline Pathogen (mMITT Analysis Set)
Description: Per pathogen microbiological response at TOC by Doripenem MIC for baseline pathogen in the mMITT analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Microbiological modified intent to treat analysis set (mMITT)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 393 | 417
Participant
  E. coli (MIC: <=0.008) - Favorable (n=1, 3) | 1 | 3
  E. coli (MIC: 0.015) - Favorable (n=160, 160) | 127 | 119
  E. coli (MIC: 0.03) - Favorable (n=112, 123) | 89 | 86
  E. coli (MIC: 0.06) - Favorable (n=14, 10) | 10 | 4
  E. coli (MIC: 0.12) - Favorable (n=3, 3) | 1 | 2
  E. coli (MIC: 0.25) - Favorable (n=1, 0) | 1 | 0
  E. coli (MIC: 0.5) - Favorable (n=0,0) | 0 | 0
  E. coli (MIC: 1) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 2) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: >16) - Favorable (n=0, 0) | 0 | 0
  Kleb.pneumoniae (MIC: <=0.008)-Favorable(n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 0.015) - Favorable (n=1, 3) | 1 | 2
  Kleb. pneumoniae (MIC: 0.03)-Favorable (n=22, 27) | 16 | 21
  Kleb. pneumoniae (MIC: 0.06)- Favorable (n=11, 16) | 10 | 7
  Kleb.pneumoniae (MIC: 0.12) -Favorable(n=4,4) | 2 | 2
  Kleb. pneumoniae (MIC: 0.25) - Favorable (n=2,3) | 1 | 2
  Kleb. pneumoniae (MIC: 0.5) - Favorable (n=2, 1) | 1 | 0
  Kleb. pneumoniae (MIC: 1) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 2) - Favorable (n= 0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 8) - Favorable (n=0, 1) | 0 | 1
  Kleb. pneumoniae (MIC: 16) - Favorable (n=0, 1) | 0 | 0
  Kleb. pneumoniae (MIC: >16) - Favorable (n=1, 0) | 1 | 0
  Proteus mirabilis (MIC:<=0.008)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.015)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.03)- Favorable (n=1, 0) | 1 | 0
  Proteus mirabilis (MIC: 0.06)- Favorable (n=2,2) | 2 | 1
  Proteus mirabilis (MIC: 0.12)- Favorable (n=6,5) | 5 | 4
  Proteus mirabilis (MIC: 0.25)- Favorable (n=6, 4) | 6 | 2
  Proteus mirabilis (MIC: 0.5)- Favorable (n=2,2) | 2 | 2
  Proteus mirabilis (MIC: 1)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 2)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 4)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 8)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 16)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: >16)- Favorable (n=0, 0) | 0 | 0
  Entero. cloacae (MIC: <=0.008)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.015)- Favorable (n= 3,1) | 2 | 1
  Entero. cloacae (MIC: 0.03)- Favorable (n= 1,5) | 1 | 2
  Entero. cloacae (MIC: 0.06)- Favorable (n= 3, 1) | 1 | 1
  Entero. cloacae (MIC: 0.12)- Favorable (n= 0, 4) | 0 | 4
  Entero. cloacae (MIC: 0.25)- Favorable (n= 0,1) | 0 | 0
  Entero. cloacae (MIC: 0.5)- Favorable (n= 4,0) | 2 | 0
  Entero. cloacae (MIC: 1)- Favorable (n= 0,1) | 0 | 1
  Entero. cloacae (MIC: 2)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 4)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 8)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 16)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: >16)- Favorable (n= 0,0) | 0 | 0
  P.aeruginosa (MIC: <=0.008) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.015) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.03) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.06) - Favorable (n=2,3) | 2 | 3
  P.aeruginosa (MIC: 0.12) - Favorable (n=2,2) | 1 | 2
  P.aeruginosa (MIC: 0.25) - Favorable (n=2,5) | 2 | 2
  P.aeruginosa (MIC: 0.5) - Favorable (n=2,1) | 2 | 1
  P.aeruginosa (MIC: 1) - Favorable (n=1,4) | 0 | 3
  P.aeruginosa (MIC: 2) - Favorable (n=1,0) | 1 | 0
  P.aeruginosa (MIC: 4) - Favorable (n=2,2) | 1 | 1
  P.aeruginosa (MIC: 8) - Favorable (n=2,1) | 1 | 1
  P.aeruginosa (MIC: 16) - Favorable (n=2,1) | 0 | 1
  P.aeruginosa (MIC: >16) - Favorable (n=2,1) | 2 | 1

56. Secondary Outcome: Per-pathogen Microbiological Response at TOC by Doripenem MIC for Baseline Pathogen (Extended ME at TOC Analysis Set)
Description: Per pathogen microbiological response at TOC by Doripenem MIC for baseline pathogen in the Extended ME at TOC analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Extended microbiological evaluable analysis set at TOC (EME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 292 | 311
Participant
  E. coli (MIC: <=0.008) - Favorable (n=1,1) | 1 | 1
  E. coli (MIC: 0.015) - Favorable (n=122, 119) | 106 | 95
  E. coli (MIC: 0.03) - Favorable (n=79, 89) | 64 | 70
  E. coli (MIC: 0.06) - Favorable (n=10, 8) | 7 | 3
  E. coli (MIC: 0.12) - Favorable (n=1, 2) | 1 | 1
  E. coli (MIC: 0.25) - Favorable (n=1, 0) | 1 | 0
  E. coli (MIC: 0.5) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 1) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 2) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: >16) - Favorable (n=0, 0) | 0 | 0
  Kleb.pneumoniae (MIC: <=0.008)-Favorable(n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 0.015) - Favorable (n=1, 2) | 1 | 1
  Kleb. pneumoniae (MIC:0.03) - Favorable (n=15, 23) | 12 | 18
  Kleb. pneumoniae (MIC: 0.06) - Favorable (n=8, 12) | 7 | 6
  Kleb.pneumoniae (MIC: 0.12) -Favorable(n=3, 2) | 2 | 2
  Kleb. pneumoniae (MIC: 0.25) - Favorable (n=2, 2) | 1 | 1
  Kleb. pneumoniae (MIC: 0.5) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 1) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 2) - Favorable (n= 0,0) | 0 | 0
  Kleb. pneumoniae (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 8) - Favorable (n=0, 1) | 0 | 1
  Kleb. pneumoniae (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: >16) - Favorable (n=1, 0) | 1 | 0
  Proteus mirabilis (MIC:<=0.008)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.015)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.03)- Favorable (n=1,0) | 1 | 0
  Proteus mirabilis (MIC: 0.06)- Favorable (n=2,2) | 2 | 1
  Proteus mirabilis (MIC: 0.12)- Favorable (n=4,2) | 4 | 2
  Proteus mirabilis (MIC: 0.25)- Favorable (n=6, 3) | 6 | 1
  Proteus mirabilis (MIC: 0.5)- Favorable (n=1,0) | 1 | 0
  Proteus mirabilis (MIC: 1)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 2)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 4)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 8)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 16)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: >16)- Favorable (n=0, 0) | 0 | 0
  Entero. cloacae (MIC: <=0.008)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.015)- Favorable (n= 1,1) | 1 | 1
  Entero. cloacae (MIC: 0.03)- Favorable (n= 1,4) | 1 | 1
  Entero. cloacae (MIC: 0.06)- Favorable (n= 2, 1) | 1 | 1
  Entero. cloacae (MIC: 0.12)- Favorable (n= 0,4) | 0 | 4
  Entero. cloacae (MIC: 0.25)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.5)- Favorable (n= 3,0) | 2 | 0
  Entero. cloacae (MIC: 1)- Favorable (n= 0,1) | 0 | 1
  Entero. cloacae (MIC: 2)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 4)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 8)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 16)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: >16)- Favorable (n= 0,0) | 0 | 0
  P.aeruginosa (MIC: <=0.008) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.015) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.03) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.06) - Favorable (n=2,3) | 2 | 3
  P.aeruginosa (MIC: 0.12) - Favorable (n=1,2) | 0 | 2
  P.aeruginosa (MIC: 0.25) - Favorable (n=2,4) | 2 | 1
  P.aeruginosa (MIC: 0.5) - Favorable (n=2,1) | 2 | 1
  P.aeruginosa (MIC: 1) - Favorable (n=1,3) | 0 | 2
  P.aeruginosa (MIC: 2) - Favorable (n=1,0) | 1 | 0
  P.aeruginosa (MIC: 4) - Favorable (n=0,2) | 0 | 1
  P.aeruginosa (MIC: 8) - Favorable (n=1,1) | 0 | 1
  P.aeruginosa (MIC: 16) - Favorable (n=2,1) | 0 | 1
  P.aeruginosa (MIC: >16) - Favorable (n=1,1) | 1 | 1

57. Secondary Outcome: Per-pathogen Microbiological Response at TOC by Doripenem MIC for Baseline Pathogen (ME at TOC Analysis Set)
Description: Per pathogen microbiological response at TOC by Doripenem MIC for baseline pathogen in the ME at TOC analysis set
Time Frame: At TOC visit. TOC visit is 21 to 25 days from Randomization
Population: Microbiological evaluable analysis set at TOC (ME at TOC)
Measure: Number; unit: Participant
Arm/Group | CAZ-AVI | Doripenem
Number analyzed (Participants) | 286 | 298
Participant
  E. coli (MIC: <=0.008) - Favorable (n=1,1) | 1 | 1
  E. coli (MIC: 0.015) - Favorable (n=122, 119) | 106 | 95
  E. coli (MIC: 0.03) - Favorable (n=79, 89) | 64 | 70
  E. coli (MIC: 0.06) - Favorable (n=10, 8) | 7 | 3
  E. coli (MIC: 0.12) - Favorable (n=1,2) | 1 | 1
  E. coli (MIC: 0.25) - Favorable (n=1,0) | 1 | 0
  E. coli (MIC: 0.5) - Favorable (n=0,0) | 0 | 0
  E. coli (MIC: 1) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 2) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  E. coli (MIC: >16) - Favorable (n=0, 0) | 0 | 0
  Kleb.pneumoniae (MIC: <=0.008)-Favorable(n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 0.015) - Favorable (n=1, 2) | 1 | 1
  Kleb. pneumoniae (MIC:0.03) - Favorable (n=15, 23) | 12 | 18
  Kleb. pneumoniae (MIC: 0.06) - Favorable (n=8, 12) | 7 | 6
  Kleb.pneumoniae (MIC: 0.12) -Favorable(n=3,2) | 2 | 2
  Kleb. pneumoniae (MIC: 0.25) - Favorable (n=2, 2) | 1 | 1
  Kleb. pneumoniae (MIC: 0.5) - Favorable (n=1,0) | 1 | 0
  Kleb. pneumoniae (MIC: 1) - Favorable (n=1, 0) | 1 | 0
  Kleb. pneumoniae (MIC: 2) - Favorable (n= 0,0) | 0 | 0
  Kleb. pneumoniae (MIC: 4) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 8) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: 16) - Favorable (n=0, 0) | 0 | 0
  Kleb. pneumoniae (MIC: >16) - Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC:<=0.008)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.015)- Favorable (n=0,0) | 0 | 0
  Proteus mirabilis (MIC: 0.03)- Favorable (n=1, 0) | 1 | 0
  Proteus mirabilis (MIC: 0.06)- Favorable (n=2,2) | 2 | 1
  Proteus mirabilis (MIC: 0.12)- Favorable (n=4,2) | 4 | 2
  Proteus mirabilis (MIC: 0.25)- Favorable (n=6, 3) | 6 | 1
  Proteus mirabilis (MIC: 0.5)- Favorable (n=1,0) | 1 | 0
  Proteus mirabilis (MIC: 1)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 2)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 4)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 8)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: 16)- Favorable (n=0, 0) | 0 | 0
  Proteus mirabilis (MIC: >16)- Favorable (n=0, 0) | 0 | 0
  Entero. cloacae (MIC: <=0.008)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.015)- Favorable (n= 1,1) | 1 | 1
  Entero. cloacae (MIC: 0.03)- Favorable (n= 1,4) | 1 | 1
  Entero. cloacae (MIC: 0.06)- Favorable (n= 2, 1) | 1 | 1
  Entero. cloacae (MIC: 0.12)- Favorable (n= 0,4) | 0 | 4
  Entero. cloacae (MIC: 0.25)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 0.5)- Favorable (n= 3,0) | 2 | 0
  Entero. cloacae (MIC: 1)- Favorable (n= 0,1) | 0 | 1
  Entero. cloacae (MIC: 2)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 4)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 8)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: 16)- Favorable (n= 0,0) | 0 | 0
  Entero. cloacae (MIC: >16)- Favorable (n= 0,0) | 0 | 0
  P.aeruginosa (MIC: <=0.008) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.015) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.03) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 0.06) - Favorable (n=2,3) | 2 | 3
  P.aeruginosa (MIC: 0.12) - Favorable (n=1,2) | 0 | 2
  P.aeruginosa (MIC: 0.25) - Favorable (n=2,4) | 2 | 1
  P.aeruginosa (MIC: 0.5) - Favorable (n=2,1) | 2 | 1
  P.aeruginosa (MIC: 1) - Favorable (n=1,3) | 0 | 2
  P.aeruginosa (MIC: 2) - Favorable (n=1,0) | 1 | 0
  P.aeruginosa (MIC: 4) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 8) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: 16) - Favorable (n=0,0) | 0 | 0
  P.aeruginosa (MIC: >16) - Favorable (n=0,0) | 0 | 0

58. Secondary Outcome: Plasma Concentrations for Ceftazidime Within 15 Minutes Before/After Dose (PK Analysis Set)
Description: Blood samples were taken on Day 3 for ceftazidime (CAZ) and avibactam (AVI) plasma concentration.
Time Frame: within 15 minutes before/after dose
Population: PK analysis set (ceftazidime within 15 minutes before/after dose)
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 480
NG/ML | 65481.2 [1260 to 3190000]

59. Secondary Outcome: Plasma Concentrations for Ceftazidime Between 30 to 90 Minutes After Dose(PK Analysis Set)
Description: Blood samples were taken on Day 3 for ceftazidime (CAZ) and avibactam (AVI) plasma concentration.
Time Frame: Between 30 to 90 minutes after dose
Population: PK analysis set (ceftazidime between 30 to 90 minutes after dose)
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 483
NG/ML | 47575.1 [749 to 414000]

60. Secondary Outcome: Plasma Concentrations for Ceftazidime Between 300 to 360 Minutes After Dose(PK Analysis Set)
Description: Blood samples were taken on Day 3 for ceftazidime (CAZ) and avibactam (AVI) plasma concentration.
Time Frame: Between 300 to 360 minutes after dose
Population: PK analysis set (ceftazidime between 300 to 360 minutes after dose)
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 481
NG/ML | 16959.6 [156 to 1640000]

61. Secondary Outcome: Plasma Concentrations for Avibactam Within 15 Minutes Before/After Dose (PK Analysis Set)
Description: Blood samples were taken on Day 3 for ceftazidime (CAZ) and avibactam (AVI) plasma concentration.
Time Frame: within 15 minutes before/after dose
Population: PK analysis set (avibactam within 15 minutes before/after dose)
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 489
NG/ML | 9307.3 [125 to 1780000]

62. Secondary Outcome: Plasma Concentrations for Avibactam Between 30 to 90 Minutes After Dose(PK Analysis Set)
Description: Blood samples were taken on Day 3 for ceftazidime (CAZ) and avibactam (AVI) plasma concentration.
Time Frame: Between 30 to 90 minutes after dose
Population: PK analysis set (avibactam between 30 to 90 minutes after dose)
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 490
NG/ML | 6587.2 [113 to 105000]

63. Secondary Outcome: Plasma Concentrations for Avibactam Between 300 to 360 Minutes After Dose(PK Analysis Set)
Description: Blood samples were taken on Day 3 for ceftazidime (CAZ) and avibactam (AVI) plasma concentration.
Time Frame: Between 300 to 360 minutes after dose
Population: PK analysis set (avibactam between 300 to 360 minutes after dose)
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 488
NG/ML | 1883.2 [26 to 336000]

ADVERSE EVENTS:
Description: The summaries for adverse events are based on the safety analysis set. There is a total of 1020 patients in safety analysis set in both protocol D4280C00002 (i.e. 517 patients) and protocol D4280C00004 (i.e. 503 patients). A total of 13 patients (out of the1033 randomized patients) did not receive any amount of IV study therapy.
Arm/Group | CAZ-AVI | Doripenem
Serious Adverse Events (participants affected / at risk) | 21/511 | 12/509
Other Adverse Events (participants affected / at risk) | 67/511 | 57/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAZ-AVI (N=511) | Doripenem (N=509)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (4) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAZ-AVI (N=511) | Doripenem (N=509)
Constipation (Gastrointestinal disorders) | 11 (11) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 6 (6)
Nausea (Gastrointestinal disorders) | 15 (16) | 10 (10)
Headache (Nervous system disorders) | 38 (41) | 40 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator submits the proposed publication and /or presentation to AZAB for review at least 60 days prior to proposed publication and/or presentation. If AZAB, requests in writing, then PI shall withhold publication and/or presentation for an additional 90 days to allow AZAB to protect its intellectual rights.